CLINICAL TRIAL: NCT03956394
Title: Takayasu Arteritis Activity Evaluation by Ultrafast Ultrasound Imaging
Acronym: TAK-UF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-02
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Takayasu Arteritis
Keywords: Cardiovascular Diseases; Vascular Diseases
MeSH Terms: conditions — Takayasu Arteritis; Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Evaluation of 10 patients with active Takayasu disease, and 10 with non-active Takayasu disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Takayasu disease (Other): UltraFast ultrasound will be performed in the usual health care, with the evaluation of carotid artery disease by Doppler ultrasound in patients hospitalized for Takayasu Arteritis Assessment.
  Interventions: Diagnostic Test: UltraFast ultrasound
- Non-active Takayasu disease (Other): UltraFast ultrasound will be performed in the usual health care, with the evaluation of carotid artery disease by Doppler ultrasound in patients hospitalized for Takayasu Arteritis Assessment.
  Interventions: Diagnostic Test: UltraFast ultrasound

INTERVENTIONS:
Diagnostic Test: UltraFast ultrasound — The patient will be hospitalized by day to perform the usual follow-up of the Takayasu disease: blood sampling and Doppler ultrasound control. Then UltraFast ultrasound doppler will be assessed.

SUMMARY:
The general activity of Takayasu vasculitis is correlated with the perfusion rate of the carotid arterial wall. This can be quantified with ultrafast ultrasound imaging in sensitive Doppler sequence associated with the concomitant injection of microbubbles (SonoVue®).

The hypothesis is that the carotid artery wall flow parameters obtained with ultrafast ultrasound imaging make possible to discriminate an active disease from an inactive disease because of the fibrous sequential arterial thickening. Thus, to improve the evaluation of Takayasu vasculitis activity and to refine the criteria for response to the various immunomodulatory treatments used.

DETAILED DESCRIPTION:
Takayasu vasculitis is a systemic inflammatory disease that causes progressive thickening and stenosis of large and medium-sized arteries (the aorta and its branches, as well as the pulmonary arteries). The classic histological aspect corresponds to a chronic inflammation localized to the arterial wall. Vascular imaging plays an important role in the diagnosis and monitoring of these patients. Although Doppler ultrasound, MRI and computed tomography can simply assess recognized inflammation criteria, such as thickening or signal intensity of the arterial wall, to recognize Takayasu vasculitis in the early stages of inflammation of the disease, there is no clear correlation between the presence of these signs and the activity or progression of the disease.

However, assessment of Takayasu vasculitis activity is difficult in daily practice because symptoms, physical examination, and biological parameters may not reliably reflect vascular inflammation. Finally, unlike other small- and medium-vessel vasculitis, histology is rarely available to diagnose and evaluate the activity of patients with Takayasu vasculitis.

In order to identify local markers of disease activity, contrast ultrasound (with injection of SonoVue® microbubbles) has shown its ability to visualize the presence of micro-vessels within the carotid wall. Ultrafast Ultrasound Imaging provides a more accurate exploration of the small vasorum vessels compared to contrast ultrasound. This technology has already been the subject of a study on cerebral microvasculature. In its application on the carotid wall, it will allow easier quantification than conventional ultrasound, by a signal analysis in ultrafast Doppler and not on the gray level, much more variable.

ELIGIBILITY:
Inclusion Criteria:

* Takayasu disease diagnosed according to the American College of Rheumatology 1990 criteria

Exclusion Criteria:

* Carotid damaged not related to Takayasu disease: atherosclerosis, post-radiation stenosis.
* Contraindication with the use of SonoVue®:

  * Unstable ischemic heart disease (recent myocardial infarction, resting angina within 7 days)
  * Acute heart failure
  * Stage III or IV heart failure
  * Severe rhythm disorders
  * Patients with right-left shunt
  * Severe pulmonary arterial hypertension (pulmonary arterial pressure> 90 mmHg)
  * Uncontrolled systemic hypertension
  * Patients with respiratory distress syndrome
  * Severe chronic obstructive pulmonary disease.
  * Acute endocarditis
  * Heart valve prostheses
  * Sepsis
  * Hypercoagulation and / or recent thromboembolic events
  * Terminal stage of kidney or liver disease.
  * Hypersensitivity to sulfur hexafluoride or any of the other ingredients of SonoVue®
* Pregnancy or breastfeeding.
* Participation in another biomedical research protocol.
* Refusal or incapacitation of language or psychic to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Quantification of the vascularity | Day 1
  Quantification of the parietal vascularization in sensitive Doppler on the common carotid artery after injection of Sonovue® contrast product: quantification of the absolute signal, relative to the carotid wall surface evaluated.

SECONDARY OUTCOMES:
Evaluate average local elasticity of the ultrafast imaging results regarding the disease activity | Day 1
  Comparison of average local elasticity by shear wave elastography (anterior and posterior walls of common carotid arteries) according to the Kerr score with ultrafast imaging results
Evaluate the carotid pulse wave velocity of the ultrafast imaging results regarding the disease activity | Day 1
  Comparison of the carotid pulse wave velocity according to the Kerr score with ultrafast imaging results
Evaluate the intima-media thickness of common carotid arteries of the ultrafast imaging results regarding the disease activity | Day 1
  Comparison of intima-media thickness of common carotid arteries (automated software) according to the Kerr score with ultrafast imaging results
Dosage of C-reactive protein | Day 1
  Evaluate relation between C-reactive protein quantity and the ultrafast imaging results
Calculation of clinical index of disease activity: Indian Takayasu Activity score 2010 (Score <2: inactive disease activity / Score ≥2 active disease activity) | Day 1
  Evaluate relation between Indian Takayasu Activity score 2010 and the ultrafast imaging results

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel MESSAS, MD, Principal Investigator — Hôpital Européen Georges-Pompidou
Locations (1):
- Hôpital Européen Georges Pompidou, Paris, France

REFERENCES:
- [Derived] Goudot G, Jimenez A, Mohamedi N, Sitruk J, Wang LZ, Khider L, Bruneval P, Messas E, Pernot M, Mirault T. Vasa vasorum interna in the carotid wall of active forms of Takayasu arteritis evidenced by ultrasound localization microscopy. Vasc Med. 2024 Jun;29(3):296-301. doi: 10.1177/1358863X241228262. Epub 2024 Mar 15. PMID 38488572